CLINICAL TRIAL: NCT06646458
Title: Xuanwu Pilot: A Prospective, Interventional, Single-arm, Before-and-after Explorative Pilot to Gain Insights on Gastrointestinal and Related Benefits of the New Senior Milk Powder
Brief Title: A Explorative Pilot Study to Gain Insights for a New Senior Milk Powder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NELN202405A
Record Dates: First submitted 2024-10-01; First posted 2024-10-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers; Healthy Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Milk Powder (study product) usage group (Experimental): Investigational Product Participants in this arm will need to take 2 times every day from baseline visit to 28 days.
  Interventions: Other: Healthy Elderly Volunteers

INTERVENTIONS:
Other: Healthy Elderly Volunteers — Take the elderly milk power 2 times every day up to 28 days

SUMMARY:
The purpose of this interventional, single-arm pilot study aimed to evaluate the new product that newly developed contains a mixture of prebiotics and probiotics to gain insights of GI function acceptance, microbiological composition and related benefits before and after study product consumption in population aged between 50-70 years.

This project also serves the purpose of formulating conceptual hypothesis and directions of exploration for future research.

The main questions it aims to answer are:

1. Microbiological change from stool samples collected at baseline and in the days after study product usage
2. Gastrointestinal function and acceptance assessed during the study period
3. Health related outcomes assessed via wearable device
4. Any safety events

No comparison group

Participants will:

1. Take study product
2. Visit the study site
3. Collect the stool sample
4. Record daily gastrointestinal tolerance and health data

ELIGIBILITY:
Inclusion Criteria:

* • Age 50-70 years (bounds included)

  * Body Mass Index (BMI) between 18.5 (bound included) and 30 (bound excluded) kg/m2.
  * Ability to comply with the protocol and assessment window:
* Product intake according to instructions.
* Willing to collect, store, deliver stool sample according to instructions.

  • Willing to adhere to instructions and restrictions during entire study period*:
* No probiotic supplementations or products supplemented with probiotics.
* No dietary fiber supplements.
* No medications may modify gastrointestinal function.

  * Fluency in speaking, reading and writing in mandarin.
  * Capability of the subject to install and use the secure study platform on the smartphone during entire study period.
  * Written informed consent. *Overruled in case of medical needs.

Exclusion Criteria:

* • Known / Existing gastrointestinal diseases or disorders diagnosed by a physician that may interfere with study.

  * Known / Existing milk protein allergies, lactose intolerance or other allergies to product ingredients.
  * Known / Existing immune diseases or disorders diagnosed by a physician that may interfere with study.
  * Use of any medication may modify gastrointestinal function: tricyclic antidepressants, SSRIs/antidepressants, opioids, ACE inhibitor, bate sympathomimetics, systemic antibiotics, intestinal antiseptics, anti-inflammatory medicines (including nonsteroidal anti-inflammatory drugs [NSAIDs] and aspirin), anti-histamines, steroids, corticosteroids, laxatives, anti-diarrhoea medication, prokinetics/dopamine-antagonists, metformin, statins, or any other stomach medication (including proton pump inhibitor [PPIs], antiacids, and antihistamine2 blockers) within 8 weeks prior to enrolment.
  * Consumption of probiotic supplementations or products supplemented with probiotics within 4 weeks prior to enrolment.
  * Subject following a special diet, including but not limited to vegan diet, ketogenic diet, low fiber diet, thickening diet etc.
  * Incapability to comply with protocol as per the judgement of the investigator.
  * Participation in any other studies involving investigational or marketed products concomitantly or 2 weeks prior to enrolment.
  * Employees and/or children/family member or relatives of employees of Danone or the participating site.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal (GI) function Questionnaire | from baseline (0 day) to the end of treatment at 28 days
  Gastrointestinal symptoms assessed the tolerance of product via the Incidence of gastrointestinal discomfort

SECONDARY OUTCOMES:
Microbiological analysis | from baseline to the end of study at 28 days
  Assess the change of intestinal bacterial distribution from stool samples collected at baseline and days after treatment compelte

OTHER OUTCOMES:
Sleep quality analysis from wearable device | from baseline (0 days) to end of treatment at 28 days
  The sleep quality collected from wearable devices changes from baseline to end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Zhang, MD, Principal Investigator — Lisheng Scientific Lab
Locations (1):
- Lisheng Scientific Lab, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No